CLINICAL TRIAL: NCT04183257
Title: Effect of Escalating Oral Vitamin D Replacement on HOMA-IR in Vitamin D Deficient Type 2 Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fawad Ahmad Randhawa, Assistant Professor of Endocrinology, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: to be ascertained
Record Dates: First submitted 2015-09-07; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Vitamin D Deficiency; Insulin Resistance; Diabetes Mellitus, Type 2
Keywords: Vitamin D; T2DM; Insulin Resistance
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D (Experimental): vitamin D arm will receive oral vitamin D in escalating dosage.
  Interventions: Drug: oral vitamin D
- Conventional (No Intervention): This arm will receive conventional treatment only.

INTERVENTIONS:
Drug: oral vitamin D — oral Vitamin D 400IU will be given and will be escalated every 2 weeks.
  Other Names: oral vitamin D 400IU
  Arms: vitamin D

SUMMARY:
In addition to its effect on maintaining calcium homeostasis and mineralization of bone, vitamin D has been linked to play a pivotal role in different medical conditions including type 2 diabetes mellitus. Vitamin D plays a major role in both insulin secretion and decreasing the insulin resistance hence has a major impact on glucose tolerance. This study is designed to determine the non-skeletal effects of vitamin D in improving the glucose tolerance in type 2 diabetic patients by decreasing the insulin resistance

DETAILED DESCRIPTION:
Pakistan stands at seventh spot amongst the world having patients suffering from Type 2 Diabetes Mellitus (T2DM) with the prevalence of approximately 6.9 million in 2007.

Among the risk factors for the development of T2DM, there is a growing evidence that deficiency of vitamin D is an independent risk factor for its development and poor glycemic control. Vitamin D plays a significant role not only in secretion of insulin from the beta cells of pancreas but it also helps in decreasing the insulin resistance at the level of target cells.

Vitamin D has received an enormous attention recently. A report from Australia indicated 1 in 3 Australians are Vitamin D deficient. Reports from Pakistan have also demonstrated Vitamin D deficiency. The study conducted by Haroon Khan et al had 562 (76.2%) females while 175 (23.8%) were males. Mean age of respondents was 36.3 years (age range 15-75 years. Females had significantly lower mean Vitamin D levels (56.2%) compared to males (15.3%).

25(OH) Vitamin D is the circulating form of vitamin D which is measurable in the blood. Vitamin D insufficiency has been defined as serum 25-hydroxyvitamin D (25(OH) D) levels below 30 ng/mL and it is common among patients with T2DM. Many studies have revealed that Vitamin D3 (calcitriol) has a role in the synthesis and the secretion of insulin by receptor mediated molecular mechanisms.

Moreover Vitamin D functions are not limited to skeletal health benefits and may extend to preservation of insulin secretion and insulin sensitivity. Studies have revealed the association between vitamin D deficiency and changes in blood glucose and insulin levels as well as sensitivity of the target tissues to insulin .Cross-sectional data provide some evidence that circulating 25-hydroxyvitamin D (25(OH) D) is inversely associated with insulin resistance, although direct measurements of insulin sensitivity are required for confirmation. Available prospective studies support a protective influence of high 25(OH) D concentrations on type 2 diabetes mellitus risk. Vitamin D receptor gene polymorphisms and vitamin D interactions with the insulin like growth factor system may further influence glucose homeostasis. The ambiguity of optimal vitamin D dosing regimens and optimal therapeutic concentrations of serum 25(OH) D limit available intervention studies.

A study found no improvement in glucose tolerance following the administration of two vitamin D doses with an interval of 2 weeks to thirty-seven non-diabetic, vitamin D-deficient adults.

Another study reported a randomised, controlled trial of vitamin D3, three fortnightly doses of 120 000 IU or placebo, in centrally obese Indian men. The subjects were not necessarily insulin resistant, but there was some improvement in postprandial insulin sensitivity following supplementation. A recent systematic review and meta-analysis on the role of vitamin D and calcium in type 2 diabetes conclude that 'there appears to be a relationship' but due to the paucity of data, an understanding of the mechanisms is incomplete.

This study has a novelty in the dosage and the frequency of administration of vitamin D which has not been studied yet. This study will enable to determine the impact of vitamin D replacement on insulin resistance in vitamin D deficient Type 2 diabetic patients and to find any correlation of serum levels of 25 hydroxyvitamin D levels with the degree of insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Age 25 to 50 years as type 2 diabetes usually diagnosed in this age range.
3. Patients having Type 2 Diabetes Mellitus
4. Taking oral antidiabetic medicines
5. Serum 25(OH) vitamin D levels below 20ng/ml having no clinical symptoms of vitamin D deficiency.
6. HOMA-IR > 2.5

Exclusion Criteria:

1. Patients having evidence of liver dysfunction and chronic renal insufficiency because it will alter the metabolism of cholecalciferol.
2. Patients having parathyroid dysfunction diagnosed on the basis of blood tests as replacement of vitamin D in these patients is very complex.
3. Patients having gastrointestinal surgeries that will alter the absorption of cholecalciferol diagnosed from detailed clinical history and clinical examination.
4. Patients having clinical features of gastroparesis diagnosed on the basis of clinical history as it can alter the absorption of vitamin D.
5. Patients having erratic control of diabetes requiring multiple hospital admissions for diabetic emergencies.
6. Pregnant and lactating mothers.

   -

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance | 3 months
  insulin resistance reduction to <2.5

SECONDARY OUTCOMES:
Glycated Hemoglobin (HbA1C) | 3 months
  Reduction by 0.5%